CLINICAL TRIAL: NCT06079567
Title: An 18-month Prospective Natural History Study to Gain Insight Into FSHD2 Pathophysiology and Disease Progression
Acronym: INSIGHT FSHD2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-PP-15
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Facioscapulohumeral Muscular Dystrophy Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- New COMs for FSHD2 patients (Experimental)
  Interventions: Diagnostic Test: Validation of new COMs for FSHD2 patients

INTERVENTIONS:
Diagnostic Test: Validation of new COMs for FSHD2 patients — Monitoring of commonly used and new COMs in FSHD2 patients

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is one of the most common inherited myopathies in adults. It is associated with genetic and epigenetic deregulation of the D4Z4 locus on the sub-telomeric region of chromosome 4q35, resulting in abnormal expression of DUX4p. Type 1 FSHD (FSHD1) is the most common form of the disease and accounts for 95% of cases, while Type 2 FSHD (FSHD2) accounts for only 5% of all FSHD cases. FSHD1 and FSHD2 are closely related in terms of genetic and epigenetic foundations, pathophysiology and clinical manifestations. Although initially described as distinct entities based on their genetics, recent information suggests that both forms of myopathy may represent the opposite ends of a spectrum of molecular diseases in which alteration of the genetic and epigenetic factors that govern DUX4 suppression in skeletal muscle have a different impact in both forms of the disease. FSHD1 and FSHD2 are both associated with re-expression of DUX4 leading to muscle atrophy, but the genetics underlying this re-expression are different, depending on whether it is type 1 or type 2. For FSHD1, it is associated with a critical contraction of the D4Z4 region and the 4qA permissive allele, leading to the expression of DUX4. In contrast, FSHD2 is caused by the inheritance of two independent genetic variations. A heterozygous mutation, mainly located on the SMCHD1 (Structural Maintenance of Chromosome flexible Hinge Domain containing 1) gene, results in a loss of function of chromatin D4Z4 repressor. This mutation, combined with the 4qA allele bearing the DU4 polyadenylation site, makes this allele permissive for the expression of the DUX4 topical gene.

Therefore, because the two forms of FSHD are genetically distinct and very few patients have FSHD2, our knowledge of the impact of chromatin D4Z4 repressors, such as SMCHD1, or the progression and severity of the disease remains very limited. It is important to note that a lack of reliable biomarkers specific to the severity and progression of the disease may prevent the development of therapies to treat patients with FSHD2. This study will allow us to better understand the natural progression of FSHD2 over time, to assess the responsiveness of clinical outcome measures (COMs) and to identify and validate inflammatory serum biomarkers predicting the severity and progression of the disease.

ELIGIBILITY:
Inclusion criteria:

* Genetically confirmed FSHD2: pathogenic mutation in SMCHD1 gene and at least one D4Z4 4qA allele;
* Age 18-75 years
* Symptomatic limb weakness
* Clinical severity score of 2 to 5 (RICCI score; range 0-5), inclusive, at screening:

  * Group ambulant patient with a RICCI score of 2 to 4
  * Group non-ambulant patient with a RICCI score of 5
* Patient giving written consent after written and oral information
* Patient affiliated to a social security system
* If taking over the counter supplements, willing to remain consistent with supplement regimen throughout the course of the study

Non inclusion criteria:

* Patients with comorbidity not related to the disease that can modify the natural evolution of the disease or would interfere with safe testing in the opinion of the Investigator
* Regular use of available muscle anabolic/catabolic agents such as corticosteroids, oral testosterone or derivatives, or oral beta agonists
* Contraindication to muscle MRI as per clinic standard practice
* Patients who has been to a tropical or subtropical country during the last 3 months
* Patients who has practiced physical exercise within 10 hours before blood test
* Patients declaring not to be fasting for at least 10 hours
* Patients following a particular diet for medical reasons and after prescription by a doctor or dietitian
* Patients who regularly consumes large quantities of alcohol
* Patients having consumed an illicit recreational drug during the last 3 months
* Patients having been vaccinated during the last 3 months
* Patients having received a blood transfusion or immunoglobulins during the last 3 months
* Patients declaring to be seropositive for HIV, HBV or HCV
* Patients having had an infectious episode during the 3 weeks preceding the visit
* Use of an experimental drug in an FSHD clinical trial within the past 30 days
* Participation in others clinical trials
* Pregnant women, breastfeeding women, women of childbearing age without contraception Pregnancy
* Patient with legal protection measures (future protection mandate, family empowerment, guardianship, curators) under Article L. 1122-2 of the French Public Health Code
* Patient refusing to participate in the study or expressing opposition to participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Minimal clinical importance of the Motor Function Measure-32 (MFM-32) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  Within MFM-32, 32 terms will be evaluated to describe patient's motor functions and grouped into 3 sub-scores at baseline and 18 months:
  D1: standing position and transfer D2: axial and proximal motor function D3: distal motor function The MFM-32 ratings rely on the use of a 4-point Likert scale based on the subject's maximal abilities without assistance (0: cannot initiate the task or maintain the starting position; 1: performs the task partially; 2: performs the task incompletely or imperfectly;3: performs the task fully and normally.)

SECONDARY OUTCOMES:
Change of the Italian Severity Score (FCS) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Italian Severity Score (FCS) ranks weakness in the face, shoulders, arms, distal, and proximal lower extremities on a 15-points scale
Change of the Clinical Severity Score (CSS) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Clinical Severity score (CSS) ranks weakness in the face, shoulders, arms, distal, and proximal lower extremities on a 10-points scale
Change of the Manual Muscle Testing (MMT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Manual Muscle Testing is a modified Medical Research Council 13-point and is used with standardized positions for each grade and each muscle following the recommendations of the FSH-DY Group. Shoulder abduction and flexion, elbow flexion and extension, wrist flexion and extension, fingers flexion and extension, hip flexion and abd/adduction, knee flexion and extension, ankle plantarflexion and dorsiflexion strength will be measured bilaterally
Change of the Hand-Held dynamometry (HHD) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  Hand-Held dynamometry (HHD) assess the isometric muscle strength in both the upper and lower limbs bilaterally (global shoulder abduction and flexion, elbow flexion and extension, hip abduction, knee extension, ankle dorsiflexion isometric strength). The required equipment is a calibrated hand-held dynamometer (MicroFet). The patient has to push against the hand-held dynamometer 3 times as hard as he can for 3-5 seconds. The maximal value will be kept for further analysis.
Change of the Pinch and Grip test from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The purpose of those tests is to measure the maximum isometric strength of the hand and forearm muscles when doing a grasping or a pinching action. The equipment required for the grip and the pinch tests is a calibrate dynamometer. The subject should be strongly encouraged to give a maximum effort. We record three trials for each hand, alternating hands with at least 30 seconds recovery between each effort. We keep the best result.
Change of the 9-Hole Peg test (9-HPT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The 9-Hole Peg Test is used to measure finger dexterity. The patient is seated at a table with a small, shallow container holding 9 pegs and a wood or plastic block containing nine empty holes. When a stopwatch is started, the patient picks up the 9 pegs one at a time as quickly as possible, puts them in the 9 holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to put the pegs and to remove them (one lap) will be recorded, 3 times alternating hands. The best trial will be registered for both hands.
Change of the repeated 9-Hole Peg test (r9-HPT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The repeated 9-Hole Peg test (r9-HPT) est a fatigability test. The same procedure like 9-HPT is repeated 5 times (5 laps) with the same hand. The total time to complete the r9-HPT is recorded and the ratio "last lap/first lap" is calculated. The patient will choose the tested hand.
Change of the classic Timed Up and Go test (classic TUG) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  Balance and mobility in patients able to walk at most 30 meters will be assessed using the classic Timed Up and Go test (TUG). The classic TUG measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk 3 meters, turn, walk back to the chair, and sit down. The best performance will be recorded.
Change of the optimized Timed Up and Go test (optimized TUG) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The optimized TUG test measures, in seconds, the time taken by patient to sit up from a lying down position (1st time interval); stand up from the mat (approximate height of 46 cm, walk 3 meters, turn, walk back to the mat, sit down (2nd time interval); and lie down to return to starting position (3rd time interval).
Change of the 6-Minute Walk Test (6MWT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The 6MWT is a measure of functional exercise capacity that requires both strength and physical endurance. It assesses how far an individual can walk in 6 minutes and has been used widely in studies of neuromuscular disease
Change of the Sit Up Test (SiUT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The SiUT measures, in seconds, the time taken by a patient to sit up from a lying down position and to return to the initial position.
Change of the repeated Sit Up Test (r-SiUT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The r-SiUT measures, in seconds, the time taken by a patient to sit up from a lying down position and to return to the initial position (1 lap). This task is repeated 5 times (5 laps). The total time to complete the trial is recorded and the ratio last lap/first lap is calculated.
Change of the Stand Up Test (SaUT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The SaUT measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm) and to return to the initial position.
Change of the repeated Stand Up Test (r-SaUT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The r-SaUT measures, in seconds, the time taken by a patient to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm) and to return to the initial position. This task is repeated 5 times (5 laps). The total time to complete the trial is recorded and the ratio last lap/first lap is calculated.
Change of the Bend Over Test (BOT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The BOT measures, in seconds, the time taken by the patient, to bend forward, knee in extension, to touch a support placed in front of the middle of the tibia and to return to the initial position
Change of the repeated Bend Over Test (r-BOT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The r-BOT measures, in seconds, the time taken by the patient, to perform 5 times consecutively the following task: to bend forward, knee in extension, to touch a support placed in front of the middle of the tibia and to return to the initial position.
Change of the Neck Flexion Fatigability Test (NFFT) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The NFFT measures, in seconds, the total time that the patient can hold the following position: in a lying position, arm relaxed on each sides of the body, the patient has to raise his head from the table flexing his neck at 45°.
Change of the respiratory function (sitting and bedside spirometry) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  Sitting and bedside spirometry allow to obtain forced vital capacity and forced respiratory volume in 1 second, two standardized outcomes commonly used to evaluate respiratory function in clinical follow up and clinical trials.
Change of the muscle composition from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  Based on T1-Dixon images, muscles will be evaluated on all available sections, and a comprehensive score describing the degree of involvement will be given between 0 (unaffected muscle) to 4 (muscle completely replaced by fatty fibrous tissue or atrophic).
  A T1-MRI score will be calculated as the sum of the scores of involvement of the individual muscles in each patient.
  Based on T2 Short T1 Inversion Recovery (STIR), muscles will be evaluated on all available sections, and a comprehensive score describing the degree of involvement was given between 0 (absence of STIR hyperintensity) and 1 (presence of area of STIR hyperintensity).
  A STIR-Magnetic Resonance Imaging (MRI) score will be calculated as the sum of the scores of involvement of the individual muscles in each patient.
Change of the score for physical function and the impact of physical limitations on daily life (PROMIS57) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The PROMIS57 is an instrument developed by the NIH PROMIS initiative. The PROMIS®-57 scales include eight items from seven primary domains: depression, anxiety, physical function, pain interference (and pain intensity), fatigue, sleep disturbance, and satisfaction with social roles. A 5-point scale is used for each instrument, except for the 0-10 pain intensity item.
  Raw scores for each of the seven short forms (domains) in PROMIS-57 are calculated, and scores are converted to T-scores for each of the seven short forms (domains) in PROMIS-57 based on the PROMIS guidelines (http:// www.healthmeasures.net).
  The T-score conversion establishes 50 as a general population mean for all PROMIS domains, and any 10-point deviation corresponds to one standard deviation (SD) difference, for easy-to-understand and consistent scoring across measures.
Change of the score for the Patient Global Impression of Change (PGIC) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The PGIC items consist of 4 questions pertaining to overall disease-related symptoms, activities of daily living, as well as mobility and respiratory issues. The items range from -3 (a great deal worse) to 0 (no change) to 3 (a great deal better)
Change of the score for the Upper Extremity Functional Index (UEFI) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Upper Extremity Functional Index (UEFI) is a validated patient reported measure for adults with upper extremity dysfunction. This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
Change of the score for the Facial Disability Index (FDI) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Facial Disability Index (FDI) is a short 5 items questionnaire which assesses the physical impact of facial weakness. The five questions are summed into total score which transformed onto a percentage scale, with 100 representing normal, and lower scores representing increasing disability.
Change of the score for the Sydney Swallow Questionnaire (SSQ) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Sydney Swallow Questionnaire (SSQ) is a 17 question, self-report inventory, which was developed to measure symptomatic severity of oral-pharyngeal dysphagia as reported by the affected patient. The questionnaire uses a 100mm long visual analogue scale (VAS) for all but one question.
Change of the score for the Swallowing Quality of Life questionnaire (SWAL-QOL) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The original SWAL-QOL scale has 44 items exploring patient's quality of life and grouped into 10 lifestyle scales:
  burden of eating difficulty; eating duration; eating desire; food selection; communication; fear; mental health; social impact; fatigue; and sleep. There is also a symptom-frequency scale in which each item is scored from 1 to 5 (1 for poorest, 5 for best quality of life). For each scale, a separate score out of 100% is calculated, with each item having the same importance. There is no global score of QOL.
Change of the score for the Multidimensional Dyspnea Profile (MDP) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The Multidimensional Dyspnea Profile (MDP) is a questionnaire which assesses overall breathing discomfort, sensory qualities, and emotional responses in laboratory and clinical settings. The MDP assesses dyspnea during a specific time or a particular activity (focus period) and is designed to examine individual items that are theoretically aligned with separate mechanisms.
Change of the FSHD-Rasch-built overall disability scale (FSHD-RODS) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The FSHD-RODS is a patient-reported disease-specific interval measure suitable for detecting activity and participation restrictions in patients with FSHD. The FSHD-RODS consists of 32 items that range in difficulty level (e.g., ability to fill in a form, ability to run). Each item is graded on an ordinal scale, with 0 representing "unable to perform", 1 representing "able to perform, but with difficulty", and 2 representing "easily performed without difficulty". A total score will be calculated based on the sum of the item scores and will range from 0-64, with a lower score representing a higher disability
Change of the fatigue severity scale (FSS) from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Change of the fall and exercise questionnaire from Baseline (V1) to 18 months (V3) | At baseline and 18 months
  A fall and exercise questionnaire will assess average monthly falls and near falls, and average weekly amount of exercise. A standard questionnaire will ask about the effect of FSHD on work/occupation.
Change of the cytokines levels in serum from Baseline (V1) to 12 months (V2) and 18 months (V3) | At baseline, 12 and 18 months
  Serum cytokines level analysis will be done using v-plex® immunoassay with the commercially available Proinflammatory Panel 1 and Cytokine Panel 1 (Meso Scale Discovery MSD). Serum cytokines level will be compared between baseline the 12-months and the 18-months follow-up.

CONTACTS AND LOCATIONS:
Locations (9):
- Leuven University, Leuven, Belgium
- France (3):
  - Nice University Hospital, Nice, Alpes M
  - APHM, Marseille, Bouches du Rhone
  - Myology Institute, Paris, Paris
- Italy (3):
  - Gemelli University Hospital, Rome, Lazio
  - Nemo Center, Milan, Lombardy
  - Pisa University, Pisa, Tuscany
- Radboud University Medical Centre Nijmegen, Nijmegen, Netherlands
- Donostia University Hospital, Donostia / San Sebastian, Guipuscoa, Spain

IPD SHARING:
Plan to Share IPD: No